CLINICAL TRIAL: NCT05873270
Title: Randomized, Controlled, Single-blind Exploratory Study of the Efficacy and Safety of Wrist and Ankle Needle Intervention on Nausea, Vomiting and Pain After Sleeve Gastric Surgery in Women
Brief Title: Randomized, Controlled, Single-blind Exploratory Study of the Efficacy and Safety of Wrist and Ankle Acupuncture Intervention on Nausea, Vomiting and Pain After Sleeve Gastric Surgery in Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: LILIAN GAO (Other)
Responsible Party: Sponsor-Investigator, LILIAN GAO, nurse, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: LGAO
Record Dates: First submitted 2023-04-10; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Laparoscopic Sleeve Gastrectomy; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
- Intervention group
  Interventions: Other: Wrist and ankle acupuncture

INTERVENTIONS:
Other: Wrist and ankle acupuncture — Patients in the intervention arm started the wrist and ankle acupuncture treatment 1 day before the surgery. Take up and down 1,2 area as a needle point, use hua tuo brand sterile acupuncture needle (specification: 0.25mm 25mm), into the skin disinfection into the needle, keep 30 subcutaneous needle and skin, when the operator under the needle, patients without acid swelling, pain, close to the skin dermis, to about 1.5 inches, give tape fixed 24h, left under the skin, until postoperative 3 day.
  Groups: Intervention group

SUMMARY:
PONV is the most common clinical presentation after surgical procedures beyond pain. A retrospective study of our center found that the postoperative incidence of LSG was 77.4%. PONV can not only cause postoperative discomfort, but also cause serious complications such as disturbance water and electrolyte balance, wound splitting, incisional hernia, and even residual gastric leakage and aspiration pneumonia, resulting in prolonged hospital stay and increased medical costs. Wrist and ankle acupuncture is a special kind of acupuncture therapy. Through subcutaneous stimulation, the electrical signal is fed back along the nerve fiber into the cerebral cortex, without dialectical treatment, and only needs the appropriate symptoms and signs of the patient. Although only in the wrist and ankle, it can solve a series of problems in the whole body, especially nausea, vomiting and pain symptoms.

DETAILED DESCRIPTION:
Patients scheduled for female sleeve gastric surgery were selected, and the trial was designed into the control group (n=33) and the intervention group (33). The intervention group was based on the control group, combined with the intervention of the wrist and ankle acupuncture, namely, the wrist and ankle acupuncture treatment was started 1 day before the surgery. Take up and down 1,2 area as a needle point, use hua tuo brand sterile acupuncture needle (specification: 0.25mm 25mm), into the skin disinfection into the needle, keep 30 subcutaneous needle and skin, when the operator under the needle, patients without acid swelling, pain, close to the skin dermis, to about 1.5 inches, give tape fixed 24h, left under the skin, until postoperative 3 day.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Guidelines for Surgical Treatment of Obesity and Type 2 Diabetes in China (2019 edition);
* ASA grades II-III; Age: 18-65 years old;
* Denial of smoking history;
* Denied any history of motion sickness or PONV;
* Female patients proposed to undergo laparoscopic sleeve gastrectomy under elective general anesthesia;
* Voluntary attended and signed informed consent.

Exclusion Criteria:

* With known drug allergies related to this study;
* Severe heart, respiratory, renal or liver diseases, and coagulation disorders;
* Psychiatric or neurological disorders;
* difficulties in communication;
* Premedication or premedical conditions limits target assessment, including use of antiemetics, opioids or corticosteroids (excluding anesthetic medication);
* Gastroesophageal reflux (GRED), clinically assessed as severe GRED or preoperative gastroscopy indicating grade B of oesophagitis or above;
* Patients undergoing combined cholecystectomy and gynecological surgery during the operation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient undergoing sleeve gastric surgery in the weight loss center of the First Affiliated Hospital of Jinan University
Study Population: Female patient undergoing sleeve gastric surgery in the weight loss center of the First Affiliated Hospital of Jinan University
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-03-23 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline pain at 24 hours after surgery | Change from Baseline pain at 24 hours after surgery
  Using Visual Analogue Scale of Pain (VASP), a score 0 represents no significant pain in the past time period; a score 1-3 represents mild pain that does not affect sleep; a score 4-6 means moderate pain that slightly affects sleep; and a score 7-10 represents severe pain leading to poor sleep or painful awakening from sleep
Change from Baseline nausea and vomitting at 24 hours after surgery | Change from Baseline nausea and vomitting at 24 hours after surgery
  PONV was scored using the Visual Nausea analog core (Visual Analog Scale of Nausea, VASN).0 represents no significant nausea and vomiting in the past period; 1-3 represents mild PONV does not affect sleep; 4-6 represents moderate PONV slightly affects sleep; and 7-10 represents severe PONV causes failed to sleep. The simplified PONV impact scale was used while performing the VASN score. The assessment of PONV severity was performed to ensure the objectivity of the outcome measures evaluation. The simplified questionnaire consisted of 2 questions, each with the corresponding score, scoring 5 points defined as clinically significant PONV

SECONDARY OUTCOMES:
Gastrointestinal function | Before discharge
  The time of first exhaust and defecation were recorded.
drug used | Before discharge
  The number, type, and duration of use of analgesic and antiemetic drugs when necessary
Quality of life situation before discharge | Before discharge
  The quality of recovery before discharge was recorded
complication | perioperative period
  The occurrence of perioperative complications was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangdong, Guangzhou, China